CLINICAL TRIAL: NCT06056076
Title: Comparison of Mini Squat and Endurance Training in Improving Quality of Life in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuro Counsel Hospital, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 344
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Endurance Training

STUDY DESIGN:
Intervention Model Description: Single blind Randomized control trial
Who Masked: Participant
Masking Description: Just participants were unaware of their intervention type
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Mini Squats at a rate of ten squats at minimum range around 10-15 degrees at start along with Interferential Therapy for 10 minutes.
  Interventions: Other: Mini Squats Training
- Group B (Active Comparator): Endurance training by the use of medium resistance therapeutic band at start along with Interferential Therapy for 10 minutes.
  Interventions: Other: Endurance Training

INTERVENTIONS:
Other: Mini Squats Training — Mini Squats at a rate of ten squats at minimum range around 10-15 degrees at start along with Interferential Therapy for 10 minutes.
  Arms: Group A
Other: Endurance Training — Endurance training by the use of medium resistance therapeutic band at start along with Interferential Therapy for 10 minutes.
  Arms: Group B

SUMMARY:
Interventional type of study in which one group of participants will be given mini squats training and other endurance training to improve the quality of life of knee osteoarthritis patients.

DETAILED DESCRIPTION:
Interventional type of study in which one group of participants will be given mini squats training and other endurance training to improve the quality of life of knee osteoarthritis patients. 3 sessions per week for 4 weeks along with interferential therapy

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* grade 2-3 OA
* No Comorbidity of serious type

Exclusion Criteria:

* Pain greater than 8 on PNS
* DM
* HTN
* Neurological conditions

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
PNS | 4 weeks
  PAin Numeric ascale with 0 means no pain and 10 means worst pain ever
SF-36 Quality of Life | 4 weeks
  Lower value means low QoL and higher value means better QoL

CONTACTS AND LOCATIONS:
Locations (1):
- Muhammad Salman, Pt, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
HAs not decided yet